CLINICAL TRIAL: NCT05099783
Title: Stepwise Strategy for Modifying Atrial Fibrillation Substrate Study - Regression of Left Atrial Fibrosis Assessed by Late Gadolinium Enhanced Magnetic Resonance Imaging
Brief Title: Stepwise Strategy for Modifying Atrial Fibrillation Substrate Study - MRI
Acronym: SAFE-MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAFE-LGEMRI
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; late gadolinium enhanced magnetic resonance imaging; atrial fibrosis
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: late gadolinium enhanced magnetic resonance imaging — Candidate inpatients or outpatients will be identified if pharmacological or electrical cardioversion has be performed and MRI were performed after cardioversion at least twice.

SUMMARY:
The investigators will conduct an observational trial, with outcome ascertainment at 3 months and 6 months after cardioversion. The primary objective is to demonstrate how cardioversion may aid in the regression of left atrial fibrosis in patients with persist atrial fibrillation as assessed by late gadolinium enhanced magnetic resonance imaging. The secondary objective is to assess the relationship between structural and functional changes with heart rhythm and heart rate.

DETAILED DESCRIPTION:
Background: Atrial fibrillation (AF) is estimated to affect over 33 million people worldwide and is associated with significant co-morbidities such as embolic stroke, heart failure, dementia. Consequently, AF poses a significant burden to the healthcare system, in both direct and indirect costs. The management of AF is complex, especially for patients with persistent AF, which is defined as sustained AF for > 7 days. It is preferable to terminate the AF and restore normal sinus rhythm for relief of symptoms associated with AF or improvement of cardiac structure and function. The maintenance of AF, especially persist AF is associated with fibrosis of left atria. Furthermore, AF itself promotes fibrosis, which in turn leads to increased conduction heterogeneity within the atrial substrate resulting in further progression of AF. In animal models, alterations in myocytes after sustained AF resemble those of myocardial hibernation. Ultimately, these structural changes would lead to Calcium overload and metabolic stress, similar changes have been observed in humans. In humans, atrial dilatation and degenerative changes have been observed. Interstitial fibrosis is the prime cause of structural remodeling in left atrium. Whether reversal of sinus rhythm can reverse fibrosis partly? The introduction of Late Gadolinium enhancement magnetic resonance imaging (LGE-MRI) sequence now allows for non-invasive and dynamic assessment of the location and extent of atrial fibrosis.

To date, no studies evaluating the regression of left atrial fibrosis after cardioversion assessed by LGE-MRI have been performed. The investigators propose to use LGE-MRI to evaluate the effects of cardioversion on atrial fibrosis. It has been shown that the extent of fibrosis can predict the success of catheter ablation procedure. For these patients with more "scar", control the progression of fibrosis and simultaneously provide respite from AF recurrence would be an extremely desirable prescription.

Objectives: To determine the regression of left atrial fibrosis in patients with persist atrial fibrillation as assessed by late gadolinium enhanced magnetic resonance imaging.

Methods: This study will be an observational trial in patients with persist AF. Candidate inpatients or outpatients will be identified if MRI were performed after pharmacological or electrical cardioversion at least twice. The heart rhythm will be assessed by medical records and telephone survey.

Objective

Primary:

The primary objective of this study is to demonstrate how cardioversion may influence the regression of left atrial fibrosis in patients with persist atrial fibrillation as assessed by LGE-MRI, using longitudinal data from a retrospective study of patients diagnosed with atrial fibrillation over a six month follow up period.

Secondary:

To study the effects of sinus rhythm in global parameters of myocardial remodeling such as right and left atrial volumes and right and left ventricular volumes.

To assess whether characteristics of MRI after cardioversion can predict the rate of atrial fibrillation sinus rhythm maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Patients carry a diagnosis of Persistent Atrial Fibrillation
* Patients have given informed consent
* Pharmacological or electrical cardioversion has be performed successfully
* late gadolinium enhanced magnetic resonance imaging (LGE-MRI) were performed after cardioversion at least twice

Exclusion Criteria:

* Prior radiofrequency ablation treatment for atrial fibrillation
* Prior cardiac surgical procedures
* Individuals with cognitive impairments who are unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidate inpatients or outpatients will be identified if pharmacological or electrical cardioversion has be performed and LGE-MRI were performed after cardioversion at least twice.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
The regression of left atrial fibrosis in patients with persist atrial fibrillation after cardioversion | 3 to 6 months
  The change in left atrial fibrosis (the core and border zone area, percentage of left atrium and segments involved) using MRI imaging, from baseline to the second measurement.

SECONDARY OUTCOMES:
The effects of sinus rhythm in global parameters of myocardial remodeling | 3 to 6 months
  The change in left atrial global parameters of MRI ( left atrial volume).
The effects of sinus rhythm in global parameters of myocardial remodeling | 3 to 6 months
  The change in left atrial parameters of echocardiography.

OTHER OUTCOMES:
The predictive value of MRI for the maintenance of sinus rhythm | 0 months
  To assess characteristics of MRI after cardioversion.

CONTACTS AND LOCATIONS:
Overall Officials: Yuehui Yin, Study Director — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thijssen VL, Ausma J, Liu GS, Allessie MA, van Eys GJ, Borgers M. Structural changes of atrial myocardium during chronic atrial fibrillation. Cardiovasc Pathol. 2000 Jan-Feb;9(1):17-28. doi: 10.1016/s1054-8807(99)00038-1. PMID 10739903
- [Background] Hobbs WJ, Fynn S, Todd DM, Wolfson P, Galloway M, Garratt CJ. Reversal of atrial electrical remodeling after cardioversion of persistent atrial fibrillation in humans. Circulation. 2000 Mar 14;101(10):1145-51. doi: 10.1161/01.cir.101.10.1145. PMID 10715261
- [Background] Marrouche NF, Wilber D, Hindricks G, Jais P, Akoum N, Marchlinski F, Kholmovski E, Burgon N, Hu N, Mont L, Deneke T, Duytschaever M, Neumann T, Mansour M, Mahnkopf C, Herweg B, Daoud E, Wissner E, Bansmann P, Brachmann J. Association of atrial tissue fibrosis identified by delayed enhancement MRI and atrial fibrillation catheter ablation: the DECAAF study. JAMA. 2014 Feb 5;311(5):498-506. doi: 10.1001/jama.2014.3. PMID 24496537